CLINICAL TRIAL: NCT06164067
Title: The Role of Cervical Consistency Index and Uterocervical Angles in Predicting Second Trimester Medical Termination
Brief Title: The Role of Cervical Consistency Index and Uterocervical Angles in Medical Termination
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: 2011-KAEK-25 2022/04-52
Record Dates: First submitted 2023-04-04; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Second Trimester Abortion; Uterocervical Angle; Cervical Consistency Index
Keywords: medical termination; uterocervical angle; abortion; second trimester
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women who abort within 24 hours: Group 1 treatment was completed in the first 24 hours ( who were completely aborted and removed the fetal material and its attachments )
  Interventions: Other: abortus within 24 hours or 24-48 hours
- Pregnant women who abort within 24- 48 hours: Group 2 consisted of patients who needed additional cycles and aborted within 24-48 hours.
  Interventions: Other: abortus within 24 hours or 24-48 hours

INTERVENTIONS:
Other: abortus within 24 hours or 24-48 hours — second trimester medical termination
  Other Names: misoprostol

SUMMARY:
The main aim of the investigator study is the success of predictivity cervical consistency index (CCI), anterior uterocervical angle (aUCA) and posterior uterocervical angle (pUCA) in second trimester terminations.

DETAILED DESCRIPTION:
This prospective clinical study includes 136 pregnant women with a diagnosis of in utero ex fetus who were hospitalized for medical termination in the gynecology service of Health Sciences University Bursa High Specialization Training and Research Hospital Gynecology and Obstetrics Clinic as a single center. The participants were divided into 2 groups as those whose treatment was completed in the first 24 hours (who were completely aborted and removed the fetal material and its attachments ) and those who aborted within 24-48 hours when additional cycles were needed. Furthermore who applied to additional treatment methods were recorded (cervical balloon, hysterotomy ) during these periods. In all pregnant women; characteristic features, abortion times, doses of misoprostol used, anterior- posterior uterocervical angle, cervical length, cervical consistency indexes and gestational weeks were saved.

ELIGIBILITY:
Inclusion Criteria:

* women who had a termination indication in the second trimester and had abortion or abortion in our hospital
* women who have had a miscarriage or abortion with a normal vaginal route or hysterotomy

Exclusion Criteria:

* multiple pregnancies
* pregnant women with misoprostol-related allergies
* scar pregnancies or heterotopic pregnancies
* patients with a history of previous conization or cervical surgery,
* patients with placental invasion anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: white people same demographics no socio- cultural difference
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
success of predictivity cervical consistency index, anterior uterocervical angle and posterior uterocervical angle | 6 months
  cervical consistency index (CCI), an ultrasound measurement that aims to estimate cervical softness by measuring the anteroposterior diameter of the uterine cervix before (AP) (millimeter) and at maximal compression (AP') with the vaginal ultrasound probe and calculating the ratio between the two measurements (AP'/AP × 100). Uterocervical angle (UCA) (degree):Transvaginal sonographic images showing technique of measurement of uterocervical angle. UCA was calculated as angle between two lines. The first line was drawn between internal (I) and external ostium (os) (E). The second line was drawn 3 cm parallel to the lower aspect of anterior inner uterine wall passing through the end of the first line at internal os. (in degrees)

SECONDARY OUTCOMES:
compare the measured ultrasonographic values | 6 months
  compare the measured ultrasonographic values with the success of predictivity cervical length.( millimeter)

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)